CLINICAL TRIAL: NCT00229541
Title: Medical In-Patient Rehabilitation in Rheumatoid Arthritis: Acceptance and Outcomes in Insurants of Compulsory Health Insurances and Statutory Pension Insurances (VERA)
Brief Title: Medical In-Patient Rehabilitation in Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: AOK Schleswig-Holstein (Industry); BEK Nord (Unknown); Draeger and Hanse BKK (Industry); DAK Gesundheit (Other); IKK Schleswig-Holstein (Unknown); TK Schleswig-Holstein (Unknown); LVA Schleswig-Holstein (Unknown); BfA (Unknown); Deutsche Rheumaliga Schleswig-Holstein (Unknown); Berufsverband Deutscher Rheumatologen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKZ 01GL0306
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2007-10-29 (Estimated); Status verified 2007-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Medical in-patient rehabilitation; Gainfully employed; Work incapacity
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IG (Experimental): intervention group, receives counselling on medical inpatient rehabilitation by statutory health insurance, is intended to apply for a 3-wek medical inpatient rehabilitation at the co-operating clinic (Bad Bramstedt)
  Interventions: Procedure: Counselling and 3-week medical in-patient rehabilitation
- KG (No Intervention): control group, receives usual care

INTERVENTIONS:
Procedure: Counselling and 3-week medical in-patient rehabilitation — Counselling and 3-week medical in-patient rehabilitation in IG
  Arms: IG

SUMMARY:
The randomised controlled trial explores the efficacy of a counselling interview on an multidisciplinary multimodal intervention to ameliorate the somatic, mental and social medical progress of rheumatoid arthritis in gainfully employed insurants of compulsory health insurances and statutory pension insurances . Additionally, the feasibility to recruit a study population via databases of compulsory health insurances is examined.

DETAILED DESCRIPTION:
Rheumatoid arthritis is the most prevalent inflammatory rheumatic disease. Limited participation of the individual patient accumulates with large amounts of indirect costs for society: About 40 % of the affected patients have to quit their jobs within the first three to four years after disease onset. Nevertheless, the German health care system still seems to lack an adequate supply, particularly in case of medical rehabilitation in early stages of disease. International clinical trials, reviews amd evidence-based guidelines emphasize the importance of an early multimodal multidisciplinary team care as in Germany provided by specialised clinics through three-week in-patient medical rehabilitation programs. The available study explores the efficacy of a counselling interview on an medical in-patient rehabilitation in a randomised controlled design. Exclusively, gainfully employed insurants of compulsory health insurances and statutory pension insurances are included in the study.

Secondary, to avoid the problem of a selection bias caused by recruitment via clinics or doctors, the RCT tests the possibility to recruit potential participants by data of the co-operating health insurances on RA-specific diagnoses of work incapacity, hospital discharge diagnoses, and medical prescriptions within the past 24 months.

Detailed process:

1. Recruitment of a potential study population via health insurance data (defined search criteria: ICD-10 diagnoses M05/06/13/79 in case of work disability/hospital discharge, RA-specific medical prescriptions within the past 24 months)
2. screening questionnaire to verify in-/exclusion criteria
3. selection of eligible insurants (RA-criteria of American College of Rheumatology, clinical expert)
4. baseline measurement (e.g. SF-36, RAQoL, FFbH-P, SPE)
5. external stratified block by block randomization: intervention group (3- week medical in-patient rehabilitation) vs. control group (usual care)
6. follow-up measurement (12 months after baseline)
7. data transfer of health insurances and pension insurances

Comparison:

Looking at a 12-months follow-up, the intervention group (3-week medical in-patient rehabilitation) is expected to show significant enhancement in somatic, mental and social medical parameters concerning rheumatoid arthritis compared to a control group receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis / psoriatic arthritis (expert decision, ACR criteria)
* Insurant of co-operating health insurance and pension insurance
* Gainfully employed
* Eligible to receive a medical in-patient rehabilitation

Exclusion Criteria:

* Polyarthritis, inflammatory intestinal diseases and diseases of connective tissue
* Currently work disabled
* Not able / not willing to co-operate
* Medical in-patient rehabilitation within past 48 months

Ages: 20 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2003-10; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
work incapacity (incidence, duration) | baseline, 12 months follow-up

SECONDARY OUTCOMES:
general health status (SF-36) | baseline, 12 months follow-up
Functional capacity (FFbH-P) | baseline, 12 months follow-up
Quality of life (RAQoL) | baseline
Subjective prognosis of gainful employment (SPE-scale) | baseline, 12 months follow-up
Somatization (SCL-90-R) | baseline, 12 months follow-up
Depression | baseline, 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Raspe, Prof.Dr.Dr., Principal Investigator — Institute for Social Medicine, University of Luebeck
Locations (1):
- Institute for Social Medicine, University of Luebeck, Lübeck, Germany

REFERENCES:
- [Result] Schlademann S, Huppe A, Raspe H. [Results of a randomised controlled trial on the acceptance and the outcomes of a counselling on medical inpatient rehabilitation in gainfully employed members of statutory health insurances with rheumatoid arthritis (clinicaltrials.gov identifier NCT00229541)]. Gesundheitswesen. 2007 Jun;69(6):325-35. doi: 10.1055/s-2007-982519. German. PMID 17642037
- See also: homepage Institute for Social Medicine, University of Luebeck — http://www.sozmed.uni-luebeck.de